CLINICAL TRIAL: NCT00376012
Title: Randomized Clinical Trial to Assess the Efficacy of Short Course Intermittent Regimens for the Treatment of HIV-Associated Tuberculosis
Brief Title: Short Course Intermittent Regimens for the Treatment of HIV-Associated Tuberculosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tuberculosis Research Centre, India (Other Government)
Responsible Party: Soumya Swaminathan, Tuberculosis Research centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: trc20A
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-05

CONDITIONS: Tuberculosis; Human Immunodeficiency Virus Infections
Keywords: Chemotherapy for TB in HIV infection
MeSH Terms: conditions — Tuberculosis | interventions — Ethambutol; Isoniazid; Rifampin; Pyrazinamide

ARMS (2):
- 1 (Active Comparator): 2EHRZ3/4RH3
  Interventions: Drug: Anti-TB drugs (Ethambutol, Isoniazid, Rifampicin and Pyrazinamide)
- 2 (Experimental): 2EHRZ3/7RH3
  Interventions: Drug: Anti-TB drugs (Ethambutol, Isoniazid, Rifampicin and Pyrazinamide)

INTERVENTIONS:
Drug: Anti-TB drugs (Ethambutol, Isoniazid, Rifampicin and Pyrazinamide) — Arm 1 is a standard six-month intermittent regimen consisting of Ethambutol, Isoniazid, Rifampicin and Pyrazinamide given thrice weekly for 2 months followed by Rifampicin and Isoniazid given thrice-weekly for 4 months.
  Arms: 1
Drug: Anti-TB drugs (Ethambutol, Isoniazid, Rifampicin and Pyrazinamide) — Arm 1 is a standard six-month intermittent regimen consisting of Ethambutol, Isoniazid, Rifampicin and Pyrazinamide given thrice weekly for 2 months followed by Rifampicin and Isoniazid given thrice-weekly for 7 months.
  Arms: 2

SUMMARY:
Title: Randomized clinical trial to assess the efficacy of short course intermittent regimens for the treatment of HIV-associated tuberculosis

Phase: Phase III trial

Population: 300 HIV positive patients with tuberculosis.

Number of Sites:Four

1. Tuberculosis Research Centre, Chennai
2. Government General Hospital, Chennai
3. Government Hospital of Thoracic Medicine, Tambaram
4. Government Rajaji Hospital, Madurai

Study Duration:36 months

Study Objective:To study the efficacy of the standard RNTCP Category I regimen (2EHRZ3 / 4RH3) the control arm vs. an extended continuation phase regimen 2EHRZ3 / 7 RH3 in the treatment of pulmonary and extrapulmonary TB in the HIV positive patients.

2. To study the relationship between stage of HIV disease and response to anti-TB treatment.

3. To study recurrences and their nature (relapse/re-infection) in detail by using RFLP analysis.

Study Design:It is a two armed prospective randomized open label controlled clinical trial with stratified random allocation based on CD4 count and sputum smear grade.

All enrolled patients will be treated according to the RNTCP guidelines during the intensive phase. In the continuation phase, Cat I patients will be stratified by CD4 counts and by smear grade, and randomly allocated either to the standard RNTCP regimen, or to an alternative extended regimen (2EHRZ3/4RH3 or 2EHRZ3/7RH3).

DETAILED DESCRIPTION:
All HIV positive patients seeking care at one of the study centers, above the age of 15 years, not suffering from a serious illness, non-pregnant and diagnosed with TB will be briefly explained the treatment trial.Patients willing to participate in the trial will be asked to provide written consent. Patients who refuse participation in the study will be managed according to the RNTCP guidelines.

All patients who provide written consent to participate in the treatment trial will be interviewed by a social worker using a standard questionnaire. Patients on anti-retroviral drugs will be excluded from the study. Blood samples will be collected from patients meeting initial eligibility criteria to test for laboratory eligibility criteria. Laboratory investigations will include complete heamogram,Renal function tests, Liver function tests, random blood sugar, urine albumin and urine sugar. Patients who fulfill laboratory criteria (hemoglobin >70 g/L, granulocyte count >1.1 X 109/L, platelet count > 100X 109/L, serum alanine amino transferase concentration <2.5 times the upper limit of normal, serum creatinine concentration <1.1mg%, random blood sugar < 140 mg/dl) will be enrolled in to the study.

Randomization and Dosing:

All patients enrolled into the treatment trial will receive supervised directly observed treatment during the intensive phase. At treatment initiation, each patient will be counseled about the importance of treatment regularity. While patients are undergoing intensive phase treatment, they will be randomized either to the standard regimen or to the extended regimen as soon as CD4 results are available. Randomization will be done according to a permuted block scheme in blocks of four, stratified by CD4 counts (> 200 and ≤200) and by smear grade (0, 1+, 2+, or 3+). The treatment assignment list will be generated before the start of trial and sequentially numbered sealed envelopes containing the treatment assigned will be prepared independently.

The treatment regimens in each arm of the trial will be as follows:

Category I RNTCP regimen 2EHRZ3/4RH3 Trial regimen 2EHRZ3/7RH3 Category II RNTCP regimen 2SEHRZ3/1EHRZ3/5EHR3 Category III RNTCP regimen 2HRZ3/4RH3. All anti-TB drugs will be administered as per the RNTCP strategy of DOTS. Patients residing in Chennai and Madurai will attend the respective centers/ sub-centers three times a week for the intensive phase of treatment (first two/three months) and then once a week during the continuation phase (four to seven months). Dosages will be as per RNTCP manual and may be modified if the patient is extremely debilitated (weight < 30 kg). Patients in all treatment arms will receive 10 mg of Pyridoxine on treatment days and Co-trimoxazole DS 1 tablet daily.

During chemotherapy, patients will be called to the clinic for monthly clinical evaluation. During follow-up visits at the clinic (monthly up to 24 months, every 3 months after that), patients will be thoroughly evaluated for likely drug toxicity and the information on adverse effects will be recorded on a standardized toxicity chart.

Compliance with therapy will be measured by checking treatment cards, DOTS provider notebooks and empty drug packets. Additionally, spot urine examination will be performed to check for acetyl isoniazid and rifampicin levels at each monthly.

Statistical analysis:

The intention-to-treat approach will be used for analyzing the data for primary and secondary end points. Annual interim analyses will be done to ensure timely identification of any significant risks or benefits to patients.

Comparisons of categorical variables will be done by chi-square test and Fisher's exact test. Continuous variables will be compared by t test or by Wilcoxon's rank sum test. Survival estimates will be made by the Kaplan-Meier method. Comparison of Kaplan-Meier survival curves will be made with the log-rank test. Multivariate analyses will be performed using Cox's proportional Hazards model.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 15 years
2. HIV positivity (on 2 different ELISA tests on the same blood sample)
3. Living in Chennai or Madurai within a defined area of intake - 25 km radius.
4. Likely to remain in the same area for at least three years after start of treatment
5. The patient is judged to be cooperative and willing for thrice-weekly attendance for the first 2/3 months and once-weekly thereafter for the next 4 to 7 months
6. Is agreeable for home visits
7. No major complications of HIV disease like encephalopathy, renal or hepatic disease or end stage disease.
8. No other medical condition that might interfere with management like diabetes, convulsions, serious cardiac disease.
9. Patients who fulfill laboratory criteria (hemoglobin =>70 g/L, granulocyte count >1.1 X 109/L, platelet count > 100X 109/L, serum alanine amino transferase concentration <2.5 times the upper limit of normal, serum creatinine concentration <1.1mg%, random blood sugar < 140 mg/dl) will be enrolled in to the study

Exclusion Criteria:

1. Resides outside area of intake.
2. Pregnancy and lactation.
3. Patients with major psychiatric illnesses and severe depression
4. Major complications of HIV disease like encephalopathy, renal or hepatic disease or end stage disease
5. Serious cardiac disease (CCF, IHD), uncontrolled diabetes mellitus, convulsions, cancer, moribund state
6. Previous antituberculosis treatment for more than 1 month.
7. Patients on ART

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2001-02; Primary Completion 2007-09 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measures are TB cure and relapse rates | 2 years

SECONDARY OUTCOMES:
Secondary Outcome measure is mortality rates. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Soumya Swaminathan, MD MNAMS, Principal Investigator — Tuberculosis Research Centre, India
Locations (1):
- Tuberculosis Research Centre, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Chaisson RE, Clermont HC, Holt EA, Cantave M, Johnson MP, Atkinson J, Davis H, Boulos R, Quinn TC, Halsey NA. Six-month supervised intermittent tuberculosis therapy in Haitian patients with and without HIV infection. Am J Respir Crit Care Med. 1996 Oct;154(4 Pt 1):1034-8. doi: 10.1164/ajrccm.154.4.8887603.
- [Background] El-Sadr WM, Perlman DC, Denning E, Matts JP, Cohn DL. A review of efficacy studies of 6-month short-course therapy for tuberculosis among patients infected with human immunodeficiency virus: differences in study outcomes. Clin Infect Dis. 2001 Feb 15;32(4):623-32. doi: 10.1086/318706. Epub 2001 Feb 9. PMID 11181127
- [Background] Perriens JH, St Louis ME, Mukadi YB, Brown C, Prignot J, Pouthier F, Portaels F, Willame JC, Mandala JK, Kaboto M, et al. Pulmonary tuberculosis in HIV-infected patients in Zaire. A controlled trial of treatment for either 6 or 12 months. N Engl J Med. 1995 Mar 23;332(12):779-84. doi: 10.1056/NEJM199503233321204. PMID 7862181
- [Background] Kassim S, Sassan-Morokro M, Ackah A, Abouya LY, Digbeu H, Yesso G, Coulibaly IM, Coulibaly D, Whitaker PJ, Doorly R, et al. Two-year follow-up of persons with HIV-1- and HIV-2-associated pulmonary tuberculosis treated with short-course chemotherapy in West Africa. AIDS. 1995 Oct;9(10):1185-91. doi: 10.1097/00002030-199510000-00011. PMID 8519456
- [Background] Alwood K, Keruly J, Moore-Rice K, Stanton DL, Chaulk CP, Chaisson RE. Effectiveness of supervised, intermittent therapy for tuberculosis in HIV-infected patients. AIDS. 1994 Aug;8(8):1103-8. doi: 10.1097/00002030-199408000-00010. PMID 7986406
- [Background] el-Sadr WM, Perlman DC, Matts JP, Nelson ET, Cohn DL, Salomon N, Olibrice M, Medard F, Chirgwin KD, Mildvan D, Jones BE, Telzak EE, Klein O, Heifets L, Hafner R. Evaluation of an intensive intermittent-induction regimen and duration of short-course treatment for human immunodeficiency virus-related pulmonary tuberculosis. Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA) and the AIDS Clinical Trials Group (ACTG). Clin Infect Dis. 1998 May;26(5):1148-58. doi: 10.1086/520275. PMID 9597244
- [Derived] Swaminathan S, Narendran G, Venkatesan P, Iliayas S, Santhanakrishnan R, Menon PA, Padmapriyadarsini C, Ramachandran R, Chinnaiyan P, Suhadev M, Sakthivel R, Narayanan PR. Efficacy of a 6-month versus 9-month intermittent treatment regimen in HIV-infected patients with tuberculosis: a randomized clinical trial. Am J Respir Crit Care Med. 2010 Apr 1;181(7):743-51. doi: 10.1164/rccm.200903-0439OC. Epub 2009 Dec 3. PMID 19965813